CLINICAL TRIAL: NCT00927589
Title: A Phase 1b, Single-arm, Open-label Clinical Trial to Evaluate Corrected QT Interval and Drug-drug Interaction of Trastuzumab on Carboplatin in the Presence of Docetaxel in Patients With Metastatic Cancer
Brief Title: A Study to Evaluate Corrected QT Interval and Drug-Drug Interaction of Trastuzumab on Carboplatin in the Presence of Docetaxel in Patients With HER2-Positive Metastatic or Locally Advanced Inoperable Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H4613g; GO01305 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Solid Cancers
Keywords: HER2+ Metastatic Cancer; HER2+ Locally Advanced Inoperable Cancer; HER2+ Solid Malignancy
MeSH Terms: interventions — Carboplatin; Docetaxel; Trastuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: carboplatin; Drug: docetaxel; Drug: trastuzumab

INTERVENTIONS:
Drug: carboplatin — Intravenous repeating dose
Drug: docetaxel — Intravenous repeating dose
Drug: trastuzumab — Intravenous repeating dose

SUMMARY:
This Phase Ib, multicenter, single-arm, open-label study is designed to evaluate the effect of trastuzumab on QTcF interval and to characterize the effects of trastuzumab on carboplatin pharmacokinetics in patients with HER2-positive metastatic or locally advanced inoperable cancer.

The QT interval is a measure of time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. The QTcF interval is the QT interval as calculated using Fridericia's correction; the QTcB interval is the QT interval as calculated using Bazett's correction.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of a HER2-positive solid malignancy in patients with metastatic or locally advanced inoperable disease
* Left ventricular ejection fraction (LVEF) >/= 50% by multiple-gated acquisition (MUGA) scan or two-dimensional echocardiography (ECHO) </= 42 days prior to Cycle 1, Day 1

Exclusion Criteria:

* History of trastuzumab treatment </= 100 days prior to Cycle 1, Day 1
* Pretreatment QTcF interval > 450 ms as determined by local assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Weber, M.D., Study Director — Genentech, Inc.
Locations (19):
- United States (19):
  - Scottsdale, Arizona
  - Beverly Hills, California
  - La Jolla, California
  - San Diego, California
  - Santa Rosa, California
  - Whittier, California
  - Miami, Florida
  - Wichita, Kansas
  - Billings, Montana
  - Farmington, New Mexico
  - The Bronx, New York
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab + Docetaxel + Carboplatin: Trastuzumab was administered at an initial dose of 6 milligrams per kilogram (mg/kg) of body weight given by intravenous (IV) infusion over 90 (±10) minutes on Cycle 1 Day 2 and Cycle 1 Day 8, followed by a maintenance dose of 6 mg/kg given by IV infusion on Day 1 of each subsequent treatment cycle (every 21 [±3] days). Docetaxel was administered as an IV dose of 75 milligrams per square meter (mg/m^2) of body surface area (BSA) on Day 1 of each study treatment cycle. Carboplatin was administered as an IV dose at a target area under the concentration-versus-time curve (AUC) of 6 milligrams per milliliter per minute (mg/mL/min) on Day 1 of each study treatment cycle. Study treatment continued until the Investigator decided to discontinue study therapy or for up to 12 months after the last participant was enrolled in the study, whichever came first.
Period: Overall Study
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Started | 59
Completed | 43 (Participants were considered to have completed the study after receiving 3 cycles of treatment.)
Not Completed | 16
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Disease Progression | 8
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Trastuzumab + Docetaxel + Carboplatin: Trastuzumab was administered at an initial dose of 6 mg/kg of body weight given by IV infusion over 90 (±10) minutes on Cycle 1 Day 2 and Cycle 1 Day 8, followed by a maintenance dose of 6 mg/kg given by IV infusion on Day 1 of each subsequent treatment cycle (every 21 [±3] days). Docetaxel was administered as an IV dose of 75 mg/m^2 of BSA on Day 1 of each study treatment cycle. Carboplatin was administered as an IV dose at a target AUC of 6 mg/mL/min on Day 1 of each study treatment cycle. Study treatment continued until the Investigator decided to discontinue study therapy or for up to 12 months after the last participant was enrolled in the study, whichever came first.
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corrected QT Interval Using Fridericia's Correction (QTcF) at Trastuzumab Steady State
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR). Trastuzumab steady state was defined as the average of the 2 ECG measurements collected on Cycle 1 Day 8 (C1D8) and Cycle 2 Day 1 (C2D1) after the trastuzumab infusion.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: ECG-evaluable participant population: received any trastuzumab, had at least 1 interpretable baseline ECG measurement recorded on C1D2 prior trastuzumab exposure, had at least 1 interpretable ECG measurement recorded on C1D8 or C2D1 corresponding to time of steady-state trastuzumab concentration, and no infusion reaction requiring drug treatments.
Measure: Mean (90% Confidence Interval); unit: milliseconds (msec)
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
milliseconds (msec) | -8.4 [-11.1 to -5.7]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Carboplatin
Time Frame: 0 to 5 minutes after end of infusion on Cycle 1 Day 1 (in absence of trastuzumab) and Cycle 2 Day 1 (in presence of trastuzumab)
Population: The pharmacokinetic (PK) analysis population for carboplatin included all participants who had a measurable ultrafiltrate or plasma carboplatin concentration at all nominal sampling time points. Participants for whom a full set of carboplatin PK samples in both Cycle 1 and Cycle 2 was not reported were excluded.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 44
Microgram per milliliter (mcg/mL)
  Cycle 1 Day 1 (in absence of trastuzumab) | 51 (15.13)
  Cycle 2 Day 1 (in presence of trastuzumab) | 52 (16.58)

3. Primary Outcome: Area Under the Curve From Time Zero to 6 Hours Post Infusion (AUC0-6hr) of Carboplatin
Description: AUC0-6hr = Area under the plasma concentration versus time curve from 0 to 6 hours post-infusion.
Time Frame: 0 to 5, 60 (±5), 120 (±10), 240 (±10), and 360 (±15) minutes after end of infusion on Cycle 1 Day 1 (in absence of trastuzumab) and Cycle 2 Day 1 (in presence of trastuzumab)
Population: The PK analysis population for carboplatin
Measure: Mean (Standard Deviation); unit: Hour*microgram/milliliter (hr*mcg/mL)
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 44
Hour*microgram/milliliter (hr*mcg/mL)
  Cycle 1 Day 1 (in absence of trastuzumab) | 115 (28.63)
  Cycle 2 Day 1 (in presence of trastuzumab) | 123 (34.99)

4. Primary Outcome: Dose-Normalized Cmax (Cmax/D) of Carboplatin
Description: Dose normalized Cmax is the maximum observed concentration of carboplatin in plasma normalized for different dose levels.
Time Frame: as for outcome 2
Population: The PK analysis population for carboplatin
Measure: Mean (Standard Deviation); unit: (mcg/mL)/(min*mg/mL)
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 44
(mcg/mL)/(min*mg/mL)
  Cycle 1 Day 1 (in absence of trastuzumab) | 9 (2.52)
  Cycle 2 Day 1 (in presence of trastuzumab) | 9 (2.76)

5. Secondary Outcome: Change From Baseline in Corrected QT Interval Using Bazett's Correction (QTcB) at Trastuzumab Steady State
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Bazette's formula (QTcB = QT divided by square root of RR). Trastuzumab steady state was defined as the average of the 2 ECG measurements collected on Cycle 1 Day 8 and Cycle 2 Day 1 after the trastuzumab infusion.
Time Frame: Baseline, Cycle 1 Day 8 and Cycle 2 Day 1
Population: ECG-evaluable participant population
Measure: Mean (90% Confidence Interval); unit: msec
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
msec | -5.9 [-9.2 to -2.6]

6. Secondary Outcome: Baseline-adjusted QTcF, QTcB, PR Interval, and QRS Duration
Description: For each postbaseline timepoint, a participant's corresponding baseline measure was subtracted from his or her average of the triplicate ECG measure to create a "baseline-adjusted" corresponding ECG measure for each participant at each postbaseline timepoint.
Time Frame: Baseline, Cycle 1 Day 2 (30 minutes postdose), Cycle 1 Day 8 (15 minutes predose), Cycle 1 Day 8 (30 minutes postdose), Cycle 2 Day 1 (15 minutes predose), and Cycle 2 Day 1 (30 minutes postdose)
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
msec
  QTcF: Cycle 1 Day 2 (30 minutes postdose) (n=49) | 3.5 (11.8)
  QTcF: Cycle 1 Day 8 (15 minutes predose) (n=50) | -9.3 (12.1)
  QTcF: Cycle 1 Day 8 (30 minutes postdose) (n=50) | -4.3 (12.0)
  QTcF: Cycle 2 Day 1 (15 minutes predose) (n=48) | -15.6 (13.3)
  QTcF: Cycle 2 Day 1 (30 minutes postdose) (n=48) | -13.4 (14.6)
  QTcB: Cycle 1 Day 2 (30 minutes postdose) (n=49) | 3.9 (9.7)
  QTcB: Cycle 1 Day 8 (15 minutes predose) (n=50) | -0.8 (14.5)
  QTcB: Cycle 1 Day 8 (30 minutes postdose) (n=50) | 1.4 (14.6)
  QTcB: Cycle 2 Day 1 (15 minutes predose) (n=48) | -13.2 (16.6)
  QTcB: Cycle 2 Day 1 (30 minutes postdose) (n=48) | -14.2 (18.6)
  PR: Cycle 1 Day 2 (30 minutes postdose) (n=49) | -0.1 (9.4)
  PR: Cycle 1 Day 8 (15 minutes predose) (n=50) | 1.4 (14.6)
  PR: Cycle 1 Day 8 (30 minutes postdose) (n=50) | 4.2 (11.8)
  PR: Cycle 2 Day 1 (15 minutes predose) (n=48) | 9.7 (13.1)
  PR: Cycle 2 Day 1 (30 minutes postdose) (n=48) | 13.7 (16.1)
  QRS: Cycle 1 Day 2 (30 minutes postdose) (n=49) | -0.1 (4.0)
  QRS: Cycle 1 Day 8 (15 minutes predose) (n=50) | -1.8 (5.5)
  QRS: Cycle 1 Day 8 (30 minutes postdose) (n=50) | -1.8 (5.8)
  QRS: Cycle 2 Day 1 (15 minutes predose) (n=48) | -0.5 (5.0)
  QRS: Cycle 2 Day 1 (30 minutes postdose) (n=48) | -0.3 (6.0)

7. Secondary Outcome: Baseline-adjusted Heart Rate
Description: For each postbaseline timepoint, a participant's corresponding baseline heart rate was subtracted from his or her average of the triplicate heart rate to create a "baseline-adjusted" corresponding heart rate for each participant at each postbaseline timepoint.
Time Frame: as for outcome 6
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
beats per minute (bpm)
  Cycle 1 Day 2 (30 minutes postdose) (n=49) | 0.5 (9.9)
  Cycle 1 Day 8 (15 minutes predose) (n=50) | 9.6 (14.9)
  Cycle 1 Day 8 (30 minutes postdose) (n=50) | 6.2 (13.7)
  Cycle 2 Day 1 (15 minutes predose) (n=48) | 3.1 (12.7)
  Cycle 2 Day 1 (30 minutes postdose) (n=48) | -0.7 (12.1)

8. Secondary Outcome: Number of Participants Within Each Absolute QTc Interval Category
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Participants with maximum QTc less than or equal to (<=) 450 msec, greater than (>) 450 to <=470 msec, >470 to <= 500 msec, or >500 msec were reported.
Time Frame: as for outcome 6
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
participants
  QTcF<=450 msec: C1D2 30 min postdose (n=49) | 44
  QTcF >450 to <=470 msec:C1D2 30min postdose (n=49) | 4
  QTcF >470 to <=500 msec: C1D2 30min postdose(n=49) | 1
  QTcF >500 msec: C1D2 30 min postdose (n=49) | 0
  QTcF<=450 msec: C1D8 15 min predose (n=50) | 49
  QTcF >450 to <=470 msec: C1D8 15 min predose(n=50) | 1
  QTcF >470 to <=500 msec: C1D8 15 min predose(n=50) | 0
  QTcF >500 msec: C1D8 15 min predose (n=50) | 0
  QTcF<=450 msec: C1D8 30 min postdose (n=50) | 48
  QTcF >450 to <=470 msec: C1D8 30min postdose(n=50) | 2
  QTcF >470 to <=500 msec: C1D8 30min postdose(n=50) | 0
  QTcF >500 msec: C1D8 30 min postdose (n=50) | 0
  QTcF<=450 msec: C2D1 15 min predose (n=48) | 48
  QTcF >450 to <=470 msec: C2D1 15 min predose(n=48) | 0
  QTcF >470 to <=500 msec: C2D1 15 min predose(n=48) | 0
  QTcF >500 msec: C2D1 15 min predose (n=48) | 0
  QTcF<=450 msec: C2D1 30 min postdose (n=48) | 48
  QTcF >450 to <=470 msec: C2D1 30min postdose(n=48) | 0
  QTcF >470 to <=500 msec: C2D1 30min postdose(n=48) | 0
  QTcF >500 msec: C2D1 30 min postdose (n=48) | 0
  QTcB<=450 msec: C1D2 30 min postdose (n=49) | 36
  QTcB >450 to <=470 msec:C1D2 30min postdose (n=49) | 10
  QTcB >470 to <=500 msec: C1D2 30min postdose(n=49) | 2
  QTcB >500 msec: C1D2 30 min postdose (n=49) | 1
  QTcB<=450 msec: C1D8 15 min predose (n=50) | 41
  QTcB >450 to <=470 msec: C1D8 15 min predose(n=50) | 7
  QTcB >470 to <=500 msec: C1D8 15 min predose(n=50) | 2
  QTcB >500 msec: C1D8 15 min predose (n=50) | 0
  QTcB<=450 msec: C1D8 30 min postdose (n=50) | 39
  QTcB >450 to <=470 msec: C1D8 30min postdose(n=50) | 9
  QTcB >470 to <=500 msec: C1D8 30min postdose(n=50) | 2
  QTcB >500 msec: C1D8 30 min postdose (n=50) | 0
  QTcB<=450 msec: C2D1 15 min predose (n=48) | 43
  QTcB >450 to <=470 msec: C2D1 15 min predose(n=48) | 4
  QTcB >470 to <=500 msec: C2D1 15 min predose(n=48) | 1
  QTcB >500 msec: C2D1 15 min predose (n=48) | 0
  QTcB<=450 msec: C2D1 30 min postdose (n=48) | 43
  QTcB >450 to <=470 msec: C2D1 30min postdose(n=48) | 5
  QTcB >470 to <=500 msec: C2D1 30min postdose(n=48) | 0
  QTcB >500 msec: C2D1 30 min postdose (n=48) | 0

9. Secondary Outcome: Number of Participants With Increase From Baseline in QTc Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Participants with maximum increase from baseline of =>30msec, 30 to <60 msec (borderline) and >=60 msec (prolonged) were summarized.
Time Frame: as for outcome 6
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
participants
  QTcF<=30 msec: C1D2 30 min postdose (n=49) | 49
  QTcF >30 to <=60 msec:C1D2 30 min postdose (n=49) | 0
  QTcF >60 msec: C1D2 30 min postdose (n=49) | 0
  QTcF<=30 msec: C1D8 15 min predose (n=50) | 50
  QTcF >30 to <=60 msec: C1D8 15 min predose (n=50) | 0
  QTcF >60 msec: C1D8 15 min predose (n=50) | 0
  QTcF<=30 msec: C1D8 30 min postdose (n=50) | 50
  QTcF >30 to <=60 msec: C1D8 30 min postdose (n=50) | 0
  QTcF >60 msec: C1D8 30 min postdose (n=50) | 0
  QTcF<=30 msec: C2D1 15 min predose (n=48) | 48
  QTcF >30 to <=60 msec: C2D1 15 min predose (n=48) | 0
  QTcF >60 msec: C2D1 15 min predose (n=48) | 0
  QTcF<=30 msec: C2D1 30 min postdose (n=48) | 48
  QTcF >30 to <=60 msec: C2D1 30min postdose (n=48) | 0
  QTcF >60 msec: C2D1 30 min postdose (n=48) | 0
  QTcB<=30 msec: C1D2 30 min postdose (n=49) | 49
  QTcB >30 to <=60 msec:C1D2 30 min postdose (n=49) | 0
  QTcB >60 msec: C1D2 30 min postdose (n=49) | 0
  QTcB<=30 msec: C1D8 15 min predose (n=50) | 50
  QTcB >30 to <=60 msec: C1D8 15 min predose (n=50) | 0
  QTcB >60 msec: C1D8 15 min predose (n=50) | 0
  QTcB<=30 msec: C1D8 30 min postdose (n=50) | 49
  QTcB >30 to <=60 msec: C1D8 30 min postdose (n=50) | 1
  QTcB >60 msec: C1D8 30 min postdose (n=50) | 0
  QTcB<=30 msec: C2D1 15 min predose (n=48) | 48
  QTcB >30 to <=60 msec: C2D1 15 min predose (n=48) | 0
  QTcB >60 msec: C2D1 15 min predose (n=48) | 0
  QTcB<=30 msec: C2D1 30 min postdose (n=48) | 48
  QTcB >30 to <=60 msec: C2D1 30min postdose (n=48) | 0
  QTcB >60 msec: C2D1 30 min postdose (n=48) | 0

10. Secondary Outcome: Number of Participants With New Abnormal U Waves on ECG
Description: The incidence of abnormal U-wave changes from baseline was determined based on centrally read ECG tracings comparing each of the three triplicate readings from the post baseline ECG time points to the baseline ECG reading. At each time point, if at least one of the three triplicate readings was abnormal, the participant was counted as abnormal for that ECG timepoint as follows: a large U wave, inverted U wave, or T-U fusion compared with baseline was considered an abnormal significant change from baseline.
Time Frame: as for outcome 6
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
participants
  C1D2 30 min postdose (n=49) | 0
  C1D8 15 min predose (n=50) | 0
  C1D8 30 min postdose (n=50) | 0
  C2D1 15 min predose (n=48) | 0
  C2D1 30 min postdose (n=48) | 0

11. Secondary Outcome: Number of Participants With New Abnormal T Waves on ECG
Description: The incidence of abnormal T-wave changes from baseline was determined based on centrally read ECG tracings comparing each of the three triplicate readings from the post baseline ECG time points to the baseline ECG reading. At each time point, if at least one of the three triplicate readings was abnormal, the participant was counted as abnormal for that ECG timepoint as follows: an inverted T, flat T, or biphasic T compared with baseline was considered an abnormal significant change from baseline. Additionally, nonspecific T-wave changes from baseline were considered as abnormal nonsignificant changes from baseline. T-wave changes from baseline due to ventricular conduction or left ventricular hypertrophy strain were considered not evaluable.
Time Frame: as for outcome 6
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
participants
  C1D2 30 min postdose (n=49) | 0
  C1D8 15 min predose (n=50) | 0
  C1D8 30 min postdose (n=50) | 0
  C2D1 15 min predose (n=48) | 0
  C2D1 30 min postdose (n=48) | 0

12. Secondary Outcome: Number of Participants With Abnormal Changes in PR Interval
Description: Criteria for abnormal changes in PR interval were defined as: =>25 percentage (%) change from baseline, an absolute value >200 msec, or >=25% change from baseline and an absolute value >200 msec.
Time Frame: as for outcome 6
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
participants
  >=25% change: C1D2 30 min postdose (n=49) | 0
  Absolute value >200msec: C1D2 30min postdose(n=49) | 2
  >=25%change and >200msec:C1D2 30min postdose(n=49) | 0
  >=25% change: C1D8 15 min predose (n=50) | 1
  Absolute value >200msec: C1D8 15 min predose(n=50) | 1
  >=25%change and >200msec: C1D8 15min predose(n=50) | 1
  >=25% change: C1D8 30 min postdose (n=50) | 0
  Absolute value >200msec: C1D8 30min postdose(n=50) | 1
  >=25%change and >200msec:C1D8 30min postdose(n=50) | 0
  >=25% change: C2D1 15 min predose (n=48) | 2
  Absolute value >200msec: C2D1 15 min predose(n=48) | 4
  >=25%change and >200msec: C2D1 15min predose(n=48) | 1
  >=25% change: C2D1 30 min postdose (n=48) | 2
  Absolute value >200msec: C2D1 30min postdose(n=48) | 4
  >=25%change and >200msec:C2D1 30min postdose(n=48) | 1

13. Secondary Outcome: Number of Participants With Abnormal Changes in QRS Interval
Description: Criteria for abnormal changes in QRS interval were defined as: >=25% change from baseline, an absolute value >110 msec, or >=25% change from baseline and an absolute value >110 msec.
Time Frame: as for outcome 6
Population: ECG-evaluable participant population. n=participants with available data at each timepoint.
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 53
participants
  >=25% change: C1D2 30 min postdose (n=49) | 0
  Absolute value >110msec: C1D2 30min postdose(n=49) | 4
  >=25%change and >110msec:C1D2 30min postdose(n=49) | 0
  >=25% change: C1D8 15 min predose (n=50) | 0
  Absolute value >110msec: C1D8 15 min predose(n=50) | 4
  >=25%change and >110msec: C1D8 15min predose(n=50) | 0
  >=25% change: C1D8 30 min postdose (n=50) | 0
  Absolute value >110msec: C1D8 30min postdose(n=50) | 4
  >=25%change and >110msec:C1D8 30min postdose(n=50 | 0
  >=25% change: C2D1 15 min predose (n=48) | 0
  Absolute value >110msec: C2D1 15 min predose(n=48) | 4
  >=25%change and >110msec: C2D1 15min predose(n=48) | 0
  >=25% change: C2D1 30 min postdose (n=48) | 0
  Absolute value >110msec: C2D1 30min postdose(n=48) | 4
  >=25%change and >110msec:C2D1 30min postdose(n=48) | 0

14. Secondary Outcome: Population Pharmacokinetics of Trastuzumab
Description: As per planned analysis, separate population pharmacokinetic analysis results are not available for the current study as this analysis is based on pooled data from multiple studies.
Time Frame: 15 (±15) minutes prior to the start of the trastuzumab infusion, and 30 (±15) minutes after the end of the infusion on Cycle 1 Day 2, Cycle 1 Day 8, Cycle 2 Day 1, and Cycle 3 Day 1
Reporting Status: Not Posted

15. Primary Outcome: Geometric Mean Ratio of Cmax/D of Carboplatin
Description: The geometric mean ratio of Cmax of carboplatin was defined as the Cmax/D of carboplatin on Cycle 1 Day 1 (in the absence of trastuzumab) divided by Cmax/D of carboplatin on Cycle 2 Day 1 (in the presence of trastuzumab).
Time Frame: as for outcome 2
Population: The PK analysis population for carboplatin
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 44
ratio | 1.02 [0.90 to 1.15]

16. Primary Outcome: Dose-Normalized AUC0-6hr (AUC0-6hr/D) of Carboplatin
Description: AUC0-6hr/D = Area under the plasma concentration versus time curve from 0 to 6 hours post-infusion, normalized by carboplatin dose level.
Time Frame: as for outcome 3
Population: The PK analysis population for carboplatin
Measure: Mean (Standard Deviation); unit: (hr*mcg/mL)/(min*mg/mL)
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 44
(hr*mcg/mL)/(min*mg/mL)
  Cycle 1 Day 1 (in absence of trastuzumab) | 19 (4.77)
  Cycle 2 Day 1 (in presence of trastuzumab) | 21 (5.83)

17. Primary Outcome: Geometric Mean Ratio of AUC0-6hr/D of Carboplatin
Description: The geometric mean ratio of AUC0-6hr/D of carboplatin was defined as the AUC0-6hr/D of carboplatin on Cycle 1 Day 1 (in the absence of trastuzumab) divided by AUC0-6hr/D of carboplatin on Cycle 2 Day 1 (in the presence of trastuzumab).
Time Frame: as for outcome 3
Population: The PK analysis population for carboplatin
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 44
ratio | 1.07 [0.96 to 1.18]

18. Primary Outcome: Plasma Decay Half-Life (t1/2) of Carboplatin
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: The PK analysis population for carboplatin. n=participants with available data at each timepoint.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 44
hr
  Cycle 1 Day 1 (in absence of trastuzumab) (n=44) | 2 (0.94)
  Cycle 2 Day 1 (in presence of trastuzumab) (n=43) | 2 (1.12)

19. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Trastuzumab
Time Frame: 30 (±15) minutes after the end of the infusion on Cycle 1 Day 2, Cycle 1 Day 8, Cycle 2 Day 1, and Cycle 3 Day 1
Population: The PK analysis population for trastuzumab included all participants who had at least 1 measurable serum trastuzumab concentration collected at a nominal sampling timepoint. Participants who did not receive a trastuzumab dose or for whom no trastuzumab PK samples were reported were excluded. n=participants with available data at each timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 57
mcg/mL
  Cycle 1 Day 2 (n=57) | 146.3 [137.3 to 155.9]
  Cycle 1 Day 8 (n=51) | 187.1 [173.1 to 202.3]
  Cycle 2 Day 1 (n=48) | 179.1 [166.8 to 192.4]
  Cycle 3 Day 1 (n=42) | 181.5 [169.5 to 194.4]

20. Primary Outcome: Minimum Observed Serum Trough Concentration (Cmin) of Trastuzumab
Time Frame: 15 (±15) minutes prior to the start of the trastuzumab infusion on Cycle 1 Day 2, Cycle 1 Day 8, Cycle 2 Day 1, and Cycle 3 Day 1
Population: PK analysis population for trastuzumab. n=participants with available data at each timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Number analyzed (Participants) | 57
mcg/mL
  Cycle 1 Day 2 (n=57) | 0.178 [0.1 to 0.2]
  Cycle 1 Day 8 (n=51) | 38.8 [30.7 to 49.2]
  Cycle 2 Day 1 (n=48) | 38.7 [32.9 to 45.5]
  Cycle 3 Day 1 (n=42) | 29.7 [24.5 to 36.1]

ADVERSE EVENTS:
Time Frame: Baseline up to study completion/early termination (28 to 42 days after the last administration of study treatment) (maximum treatment duration = 163 weeks)
Description: The safety-evaluable participant analysis population included all participants who were treated with at least one dose of any treatment of the study regimen.
Arm/Group | Trastuzumab + Docetaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 26/58
Other Adverse Events (participants affected / at risk) | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Docetaxel + Carboplatin (N=58)
Small intestinal obstruction (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal spasm (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 3
Clostridium difficile colitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Haemoglobin decreased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Electrical burn (Injury, poisoning and procedural complications) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Docetaxel + Carboplatin (N=58)
Neutrophil count decreased (Investigations) | 37
Haemoglobin decreased (Investigations) | 33
Platelet count decreased (Investigations) | 23
White blood cell count decreased (Investigations) | 16
Weight decreased (Investigations) | 7
Electrocardiogram QT prolonged (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 3
Gamma- glutamyltransferase increased (Investigations) | 3
Nausea (Gastrointestinal disorders) | 34
Diarrhoea (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 31
Pyrexia (General disorders) | 13
Oedema peripheral (General disorders) | 10
Pain (General disorders) | 5
Chills (General disorders) | 4
Chest discomfort (General disorders) | 3
Mucosal inflammation (General disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 14
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hyponatraemia (Metabolism and nutrition disorders) | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Iron deficiency (Metabolism and nutrition disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 13
Dizziness (Nervous system disorders) | 12
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 18
Rash (Skin and subcutaneous tissue disorders) | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Urinary tract infection (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Candidiasis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Hypotension (Vascular disorders) | 6
Deep vein thrombosis (Vascular disorders) | 4
Flushing (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Lacrimation increased (Eye disorders) | 9
Vision blurred (Eye disorders) | 6
Insomnia (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Haematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Lymphopenia (Blood and lymphatic system disorders) | 4
Drug hypersensitivity (Immune system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.